CLINICAL TRIAL: NCT01615380
Title: Using a YMCA Exercise Program to Enhance Nicotine Dependence Treatment for Women
Brief Title: Exercise to Enhance Smoking Cessation for Women at the YMCA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA021729 (NIH); R01DA021729 (NIH)
Record Dates: First submitted 2012-05-18; First posted 2012-06-08 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Smoking
Keywords: smoking cessation; Aerobic Exercise; Women; YMCA
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT+ Contact (Active Comparator): In addition to the smoking cessation program, those in the CBT + CONTACT condition will enroll in a Wellness Program and will receive weekly wellness materials to read as well as receiving 4 sessions with a health educator in weeks 1, 4, 8 and 12 to discuss the wellness materials.
  Interventions: Behavioral: CBT+ Contact
- CBT+ Exercise (Experimental): Participants will receive an identical 12-week cognitive behavioral smoking cessation program delivered by YMCA staff and monitored by members of the research team to ensure fidelity of treatment delivery. In addition to the smoking cessation program, those in the CBT + EXERCISE condition will enroll in the 12-week YMCA Personal Fitness Program (PFP) where they will receive 4 sessions with a personal trainer in weeks 1, 4, 8 and 12 and will engage in aerobic exercise at least 3 times per week either in the PFP facilities or in other programs offered at the YMCA, such as aerobics classes.
  Interventions: Behavioral: CBT+ Exercise

INTERVENTIONS:
Behavioral: CBT+ Contact — In addition to the smoking cessation program, those in the CBT + CONTACT condition will enroll in a Wellness Program and will receive weekly wellness materials to read as well as receiving 4 sessions with a health educator in weeks 1, 4, 8 and 12 to discuss the wellness materials.
  Arms: CBT+ Contact
Behavioral: CBT+ Exercise — Participants will receive an identical 12-week cognitive behavioral smoking cessation program delivered by YMCA staff and monitored by members of the research team to ensure fidelity of treatment delivery. In addition to the smoking cessation program, those in the CBT + EXERCISE condition will enroll in the 12-week YMCA Personal Fitness Program (PFP) where they will receive 4 sessions with a personal trainer in weeks 1, 4, 8 and 12 and will engage in aerobic exercise at least 3 times per week either in the PFP facilities or in other programs offered at the YMCA, such as aerobics classes.
  Arms: CBT+ Exercise

SUMMARY:
Approximately 21% of women continue to smoke cigarettes despite the increased risk of cancer and cardiovascular disease associated with cigarette smoking. Exercise has been shown to be an efficacious treatment component in combating nicotine dependence, especially among women for whom concerns about weight gain during smoking cessation are an obstacle to successful quitting. In previous trials of women smokers, the investigators program of cognitive behavioral smoking cessation treatment (CBT) plus regular aerobic exercise was more efficacious than CBT plus equal contact time. Recognizing the program's successes, Commit to Quit (CTQ) was recently designated an Effective Program by the Substance Abuse and Mental Health Services Administration's (SAMHSA) National Registry of Effective Programs. Thus, the Commit to Quit program is well poised for a larger trial in a community setting where it has the potential to reach a large number of female smokers in a setting in which it can be sustained. In response to PA-03-126, Behavioral Therapies Development Program, the investigators propose a Stage III study in which they will conduct a trial to test the investigators CTQ smoking cessation program in the community setting of the local YMCAs. As stated in the PA, Stage III research is aimed at understanding if and how an efficacious therapy may be transported to the community. The investigators propose a randomized controlled clinical trial to take place in the YMCA setting and delivered by YMCA staff. The trial will compare CBT smoking cessation treatment plus a program of regular exercise to CBT smoking cessation treatment plus contact control. In order to promote transportability to the YMCA, the investigators will use the YMCA's existing Personal Fitness Program, which is similar to the investigators CTQ exercise program, in that it is guided by trained staff and requires participants to exercise 3 times per week. If the exercise condition is found to be more efficacious than contact control when delivered at the YMCA by YMCA staff, then the investigators will be well positioned to partner with the YMCA to pursue widespread, national dissemination of this program.

DETAILED DESCRIPTION:
We propose a randomized controlled clinical trial to take place in the YMCA setting and to be delivered by YMCA staff. The trial will compare CBT smoking cessation treatment plus a program of regular exercise (CBT + EXERCISE) to CBT smoking cessation treatment plus an equal staff contact control (CBT + CONTACT). In order to promote transportability to the YMCA, the exercise program will be the YMCA's existing Personal Fitness Program, which like our CTQ exercise program, is guided by trained staff and requires participants to exercise at least 3 times per week.

If CBT + EXERCISE is found to be more efficacious than CBT + CONTACT when delivered at the YMCA by YMCA staff, then we will be well positioned to partner with the YMCA's initiative of Y Total Health to pursue widespread, national dissemination of this program. The proposed testing of the efficacy of the CTQ program in the YMCA setting is a necessary intermediate step in the eventual dissemination of the CTQ program.

Primary Aim. To determine the efficacy of CBT + EXERCISE compared with CBT + CONTACT when delivered in the YMCAs by YMCA staff to enhance the achievement and maintenance (3, 6, and 12 months follow-up) of smoking cessation (continuous abstinence) among healthy adult female smokers.

Hypothesis. Participants in the CBT + EXERCISE condition will have significantly greater continuous abstinence rates than those in the CBT + CONTACT condition at end-of-treatment, 3, 6, and 12 months follow-up.

Additional Questions of Interest.

1. To perform process-to-outcome analyses on the intermediate variables which influence the achievement and maintenance of smoking cessation among healthy female smokers. Specifically, to determine if exercise affects weight and/or weight concerns, negative affect associated with nicotine withdrawal, and/or self-efficacy and to determine if these hypothesized mediators affect the achievement and maintenance of smoking cessation.

To explore potential moderators of the treatment, such as baseline demographic and psychological characteristics (e.g., age, baseline mood) on smoking cessation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female smokers
* ages 18 - 65
* Read and write English
* Regularly smoke 5 or more cigarettes a day
* Sedentary, or not exercising greater than 20 minutes of vigorous exercise more than once a week or greater than 30 minutes of moderate exercise 2 times per week.

Exclusion Criteria:

* known history of cardiovascular
* pulmonary or metabolic disease such as coronary artery disease, stroke, hypertension, chronic bronchitis, asthma, emphysema, and diabetes
* Any musculoskeletal problems that would limit exercise training such as knee or hip osteoarthritis or any other serious medical condition that might make exercise unsafe or unwise.
* The current use of smokeless tobacco, nicotine replacement therapy or other smoking cessation treatment, and currently using prescription medication that might impair exercise performance or tolerance, specifically beta-blockers or medications used for the treatment of hypertension
* Pregnant or planning to become pregnant within the next 12 months.
* Women hospitalized for a psychiatric disorder
* Receiving treatment for bipolar disorder or schizophrenia
* Current alcohol abuse or psychological problems when quitting in the past that required treatment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2006-09; Primary Completion 2010-09 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Salivary Cotinine | 12 months posttreatment
  Saliva will be collected at the 12 month follow-up visit and sent to a laboratory for analysis of cotinine, a biomarker of nicotine.

CONTACTS AND LOCATIONS:
Overall Officials: Bess H Marcus, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Mriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Whiteley JA, Williams DM, Dunsiger S, Jennings EG, Ciccolo JT, Bock BC, Albrecht A, Parisi A, Linke SE, Marcus BH. YMCA commit to quit: randomized trial outcomes. Am J Prev Med. 2012 Sep;43(3):256-62. doi: 10.1016/j.amepre.2012.05.025. PMID 22898118